CLINICAL TRIAL: NCT04119427
Title: The Safety and Efficacy of Micro-energy Ultrasound in the Treatment of Renal Insufficiency After Renal Transplantation: A Multicenter, Randomized Clinical Trail
Brief Title: The Safety and Efficacy of Micro-energy Ultrasound in the Treatment of Renal Insufficiency After Renal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-194
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Renal Insufficiency; Renal Transplantation
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): After installing the disposable treatment head coat, the transplanted kidney was treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed. Patients were treated twice a week for 6 weeks.
  Interventions: Device: ultrasonic therapeutic apparatus 1
- Control Group (Placebo Comparator): The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.
  Interventions: Device: ultrasonic therapeutic apparatus 2

INTERVENTIONS:
Device: ultrasonic therapeutic apparatus 1 — After installing the disposable treatment head coat, the transplanted kidney was treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed. Patients were treated twice a week for 6 weeks.
  Arms: Test Group
Device: ultrasonic therapeutic apparatus 2 — The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.
  Arms: Control Group

SUMMARY:
The safety and efficacy of micro-energy ultrasound in the treatment of renal insufficiency after renal transplantation.

DETAILED DESCRIPTION:
1. Study purposes: To evaluate the safety and efficacy of micro-energy ultrasound in the treatment of renal dysfunction after renal transplantation by measuring serum creatinine, urine volume, urea nitrogen, and transplanted kidney ultrasound, etc.
2. Study design: This is a randomized, double-blind, controlled, multicenter clinical trial.
3. Study objects: Patients with mild to moderate renal insufficiency after renal transplantation.
4. Number of samples: 90
5. Main study center: Department of Urology, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China.
6. Treatments:

Test group: After installing the disposable treatment head coat, the transplanted kidney was treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed.Patients were treated twice a week for 6 weeks.

Control group: The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.

ELIGIBILITY:
Inclusion Criteria:

1. More than half a year after renal transplantation, serum creatinine elevated over three times , patients with ineffective immunosuppressive drugs;
2. Mild to moderate renal insufficiency (creatinine less than 442umol / L);
3. Volunteer to participate in this clinical trial, comply with the requirements of this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Patients with severe renal insufficiency;
2. Blood routine suggests acute and chronic blood system diseases;
3. B-ultrasound suggests transplanting hydronephrosis;
4. Uncontrollable patients with diabetes, hypertension, and cardiovascular disease;
5. The investigator determined that it is not suitable for this clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring the patient'serum creatinine by a biochemical analyzer | within 3 months after surgery
  Measuring the patient'serum creatinine by a biochemical analyzer
Manually record the patient's urine volume in 24 hours by a measuring glass | within 3 months after surgery
  Manually record the patient's urine volume in 24 hours by a measuring glass
Measuring the patient'urea nitrogen by a biochemical analyzer | within 3 months after surgery
  Measuring the patient'urea nitrogen by a biochemical analyzer

SECONDARY OUTCOMES:
Monitoring the blood flow of the transplanted kidney by a doppler ultrasound | within 3 months after surgery
  Monitoring the blood flow of the transplanted kidney by a doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China